CLINICAL TRIAL: NCT06254300
Title: Online Exercise Program During Perioperative Treatment in Adults With Gastric Cancer (On4Cancer): Randomized Controlled Trial
Brief Title: Online Exercise Program During Perioperative Treatment in Adults With Gastric Cancer
Acronym: On4Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maia (Other)
Responsible Party: Principal Investigator, Lia Bahut, Principal Investigator, University of Maia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: On4Cancer
Record Dates: First submitted 2024-01-23; First posted 2024-02-12 (Actual); Last update posted 2024-02-12 (Actual); Status verified 2024-02

CONDITIONS: Gastric Cancer
Keywords: Physical Exercise; Gastric Cancer; Prehabilitation; Perioperative Cancer Treatment
MeSH Terms: conditions — Stomach Neoplasms; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): The intervention group will participate in a supervised online exercise prehabilitation program that will extend throughout the chemotherapy until one week before the scheduled surgery. The exercise program will consist of three sessions per week, each lasting 60 minutes. The design of the prehabilitation program is based on exercise prescription recommendations for cancer survivors and will be tailored to each patient's initial functional capacity. The exercise sessions will be conducted at home through an online platform, enabling real-time interaction among groups of patients.
  Interventions: Behavioral: Exercise Training
- Control Group (No Intervention): Participants from the control group will be offered optimal medical care, which includes general advice about healthy lifestyle including regular physical activity participation according to the current guidelines.

INTERVENTIONS:
Behavioral: Exercise Training — The exercise program will consist of three sessions per week, each lasting 60 minutes. The aerobic exercise will gradually increase the duration throughout the program to 40 minutes and exercise intensity from 30% to 59% of heart rate reserve. The resistance training will include bodyweight functional exercises and resistance exercises using elastic bands. The intensity of resistance exercise will progressively increase according to levels of progressive length and resistance of the elastic bands. The volume of resistance training will start with one set of 8 repetions. It will then gradually increase alongside the program to 2 sets of 12 repetitions. Participants will also be guided to assess their subjective effort using the Borg scale (RPE 12-15).
  Arms: Intervention Group

SUMMARY:
Perioperative chemotherapy with fluorouracil, leucovorin, oxaliplatin, and docetaxel (FLOT4) is the standard perioperative treatment for resectable and advanced gastric adenocarcinoma. Although the FLOT4 regimen have shown increases in the overall survival, response rate, and progression-free survival, it is also associated with substantial toxicities. Prehabilitation is an effective strategy to improve physical fitness in cancer patients and reverse functional limitations and inadequate levels of physical activity that are associated with worse postoperative outcomes and treatment response. Therefore, the main objective of this study is to evaluate the effects of an online, supervised exercise-based prehabilitation program on the cardiorespiratory fitness level, functional fitness and quality of life among adults with gastric cancer undergoing neoadjuvant chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Willingness to participate in the study.
* Referral for surgical treatment for gastric cancer.
* Diagnosis of gastric cancer for curative intent - stage II/III
* Referall to the perioperative FLOT4 chemotherapy regimen
* ECOG PS 0-1.
* Receptiveness and availability to use the proposed technology for exercise sessions

Exclusion Criteria:

* Inability to provide informed consent
* Inability to engage in physical training or perform the baseline walking test
* Presence of distant metastatic disease
* History of previous or concurrent malignancy
* Diagnosis of heart failure, ischemic heart disease, or sinus node valvular disease
* Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-03-23 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Aerobic capacity | Change from baseline to 1 week before surgery
  Incremental Shuttle Walk Test (ISWT)

SECONDARY OUTCOMES:
Aerobic capacity | Change from 1 week before surgery to 30 days post-surgery
  Incremental Shuttle Walk Test (ISWT)
Aerobic capacity | Change from 30 days post-surgery to 15 days after the conclusion of curative treatment
  Incremental Shuttle Walk Test (ISWT)
Muscle strength | Change from baseline to 1 week before surgery
  Digital hand dynamometer
Muscle strength | Change from 1 week before surgery to 30 days post-surgery
  Digital hand dynamometer
Muscle strength | Change from 30 days post-surgery to 15 days after the conclusion of curative treatment
  Digital hand dynamometer
Body composition | Change from baseline to 1 week before surgery
  Bioelectrical impedance
Body composition | Change from 1 week before surgery to 30 days post-surgery
  Bioelectrical impedance
Body composition | Change from 30 days post-surgery to 15 days after the conclusion of curative treatment
  Bioelectrical impedance
Health-related quality of life | Change from baseline to 1 week before surgery
  European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30). The final scores will range from 0 to 100, with higher scores on the functional scales representing a high level of functioning and higher scores on the symptom scales implying a stronger symptom burden.
Health-related quality of life | Change from 1 week before surgery to 30 days post-surgery
  European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30). The final scores will range from 0 to 100, with higher scores on the functional scales representing a high level of functioning and higher scores on the symptom scales implying a stronger symptom burden.
Health-related quality of life | Change from 30 days post-surgery to 15 days after the conclusion of curative treatment
  European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30). The final scores will range from 0 to 100, with higher scores on the functional scales representing a high level of functioning and higher scores on the symptom scales implying a stronger symptom burden.
Gastric cancer specific health-related quality of life | Change from baseline to 1 week before surgery
  The European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire-Stomach (EORTC QLQ-STO22). The final scores will range from 0 to 100, with higher scores indicating worse symptomatic problems.
Gastric cancer specific health-related quality of life | Change from1 week before surgery to 30 days post-surgery
  The European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire-Stomach (EORTC QLQ-STO22). The final scores will range from 0 to 100, with higher scores indicating worse symptomatic problems.
Gastric cancer specific health-related quality of life | Change from 30 days post-surgery to 15 days after the conclusion of curative treatment
  The European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire-Stomach (EORTC QLQ-STO22). The final scores will range from 0 to 100, with higher scores indicating worse symptomatic problems.
Physical activity | Change from baseline to 1 week before surgery
  Accelerometer (wGT3X, ActiGraph LLC, Pensacola, FL, USA)
Physical activity | Change from 1 week before surgery to 30 days post-surgery
  Accelerometer (wGT3X, ActiGraph LLC, Pensacola, FL, USA)
Physical activity | Change from 30 days post-surgery to 15 days after the conclusion of curative treatment
  Accelerometer (wGT3X, ActiGraph LLC, Pensacola, FL, USA)
Calf circumference | Change from baseline to 1 week before surgery
Calf circumference | Change from 1 week before surgery to 30 days post-surgery
Calf circumference | Change from 30 days post-surgery to 15 days after the conclusion of curative treatment
Postoperative morbidity outcomes | Within 30 days after surgery
  Clavien-Dindo classification
Treatment compliance | Through chemotherapy completion
  Relative dose intensity, calculated as the ratio of the delivered dose intensity to the standard dose intensity
Adverse events | During the treatment (neoadjuvant chemotherapy)
  Patient-Reported Outcomes Version of the Common Terminology Criteria for Adverse Events (PRO-CTCAE)
Number of hospitalizations | Within 30 days after surgery
Length of hospital stay | Within 30 days after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Centro Hospitalar de Vila Nova de Gaia/Espinho, Vila Nova de Gaia, Portugal

IPD SHARING:
Plan to Share IPD: Yes